CLINICAL TRIAL: NCT05632783
Title: A Phase 3, Multicenter, Randomized, Double-blind Study to Evaluate the Efficacy, Safety, and Tolerability of Chondroitin Sulfate 800 mg Tablets Versus Placebo in Subjects With Pain Due to Knee Osteoarthritis and to Evaluate the Durability of the Effect and Safety of the Treatment
Brief Title: TreatMent Of Knee osTeoarthritis wIth chONdroitin Sulfate - the OA MOTION Study
Acronym: MOTION
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study canceled before starting
Sponsor: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22US-Ct04
Record Dates: First submitted 2022-11-17; First posted 2022-12-01 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2022-11

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Chondroitin Sulfates

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study. Matching placebo tablets, indistinguishable from the test drug 800 mg chondroitin sulfate tablets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- chondroitin sulfate 800 mg tablets (Experimental): oral chondroitin sulfate 800 mg tablet
  Interventions: Drug: Chondroitin Sulfate Sodium
- placebo (Placebo Comparator): oral placebo tablets matching the IP tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Chondroitin Sulfate Sodium — Chondroitin sulfate 800 mg tablets
  Other Names: chondroitin sulfate 800 mg
  Arms: chondroitin sulfate 800 mg tablets
Other: Placebo — Placebo tablets
  Arms: placebo

SUMMARY:
The goal of this phase III study is to evaluate the efficacy, safety, and tolerability of chondroitin sulfate 800 mg oral tablets versus placebo in the treatment of subjects with pain due to knee OA (osteoarthritis). The further aims of the study are to evaluate the durability of the treatment effect (up to week 36) and to gain further long-term safety and efficacy data (up to 48 weeks).

The primary outcome of interest will be the effect of chondroitin sulfate on pain in the index knee at week 24 compared to placebo.

The effect of chondroitin sulfate in the index knee functionality and the patient global impression of changes at 24 weeks compared to placebo are included as key-secondary endpoints. An additional key secondary endpoint will assess the durability of the effect on pain compared to placebo at week 36. Several additional secondary endpoints are included to further support the beneficial effect of the treatment and the improvements in patient's quality of life (i.e., Western Ontario and McMaster Universities Arthritis Index -WOMAC- subscales and total scores at each study visits, changes in patient's quality of life, use of rescue medication etc.) other than the safety of the product.

DETAILED DESCRIPTION:
The goal of this phase III study is to evaluate the efficacy, safety, and tolerability of chondroitin sulfate 800 mg oral tablets versus placebo in the treatment of subjects with pain due to knee OA (osteoarthritis). The further aims of the study are to evaluate the durability of the treatment effect (up to week 36) and to gain further long-term safety and efficacy data (up to 48 weeks). Approximately 690 male and female adult subjects with moderate-to-severe pain due to OA of the knee will be randomized in a 1:1 ratio to receive either chondroitin sulfate 800 mg tablets (CS) or matching placebo. Subjects will orally self administer chondroitin sulfate/placebo once daily at home during the double blind treatment period of 36 weeks. The first approximately 250 subjects who reach Week 36 and are willing to further participate in the study will attend a double blind long-term safety follow-up period and will continue to self administer chondroitin sulfate/placebo for 12 additional weeks (up to week48). Acetaminophen 500 mg oral tablets, max. 6 tablets per day (rescue medication), will be the only analgesic allowed for the clinical study to treat pain of any type.

The study will include the following endpoints:

Primary Efficacy (Double-blind Treatment Period until Week 36) • Change from Baseline to Week 24 in the weekly mean of the average daily pain in the index knee as measured by the numerical rating scale (NRS) (0 10 points)

Key Secondary Efficacy (Double-blind Treatment Period until Week 36)

* Change from Baseline to Week 24 in Western Ontario and McMaster Universities Arthritis Index (WOMAC) function subscale
* Subject's global evaluation at Week 24 as measured by Patient Global Impression of Change (PGIC)
* Change from Baseline to Week 36 in the weekly mean of the average daily pain in the index knee as measured with the NRS (durability of effect)

Other Secondary Efficacy (Double-blind Treatment Period until Week 36)

* Change from Baseline to each week until Week 36 in the weekly mean of the average daily pain in the index knee as measured with the NRS
* Change from Baseline to Weeks 4, 12, 24, and 36 in WOMAC total score and all WOMAC subscores
* Consumption of rescue medication (acetaminophen), including the number of intake days, number of daily intakes, and total dose per day
* Change from Baseline to Weeks 4, 12, 24, and 36 in subject's quality of life (Short Form 36 Health Survey Questionnaire [SF-36])
* Subject's global evaluation at Weeks 4, 12, and 36 as measured by PGIC
* Investigator's global evaluation at Weeks 4, 12, 24, and 36 by Clinician Global Impression of Change (CGIC)
* Responder rates at each visit using 2 different response definitions (≥30% or ≥50% decrease in weekly mean of the average daily [24 hour] NRS pain intensity score)

Safety and Tolerability (Double-blind Treatment Period until Week 36)

* Number of subjects with any adverse events (AEs), treatment emergent adverse events (TEAEs), AEs causally related to the investigational product (IP) (ADRs), and serious adverse events (SAEs)
* Number of dropouts due to AEs and dropouts due to AEs causally related to the IP (ADRs)
* IP Compliance
* Subject's treatment satisfaction as measured by the Medication Satisfaction Questionnaire (MSQ) at Weeks 4, 12, 24, and 36
* Change in laboratory parameters from Baseline to Weeks 4, 12, 24, and 36
* Change in 12 lead electrocardiogram (ECG) parameters from Baseline to Week 24
* Change in vital signs from Baseline to each post-baseline visit

Safety Follow-up Period from Weeks 36 to 48 with Continued Double-blind Treatment for those subjects who continue in the study until Week 48 (planned number: approximately 250 subjects)

Primary Safety

• Number of subjects with any AEs, TEAEs, ADRs, and SAEs

Secondary Safety

* Changes from Baseline to Week 48 in vital signs, ECG, and safety laboratory results
* Changes from Baseline to Week 48 in subject's treatment satisfaction as measured by the MSQ

Exploratory Efficacy

* To explore the long-term efficacy of once daily treatment with CS 800 mg oral tablets
* Change from Baseline to Week 48 in the weekly mean of the average daily pain in the index knee as measured by the NRS (0 10 points)
* Change from Baseline to Week 48 in WOMAC total score and all subscale scores
* Change from Baseline to Week 48 in subject's quality of life (SF-36)
* Subject's global evaluation as measured by PGIC at Week 48
* Investigator's global evaluation as measured by CGIC at Week 48

Subjects will use an eDiary (electronic diary) to record, daily, their average daily pain in the index knee (by a numerical rating scale) and to record the daily administration of the IP and the frequency and dose of rescue medication taken.

To enter the study, subjects must be outpatients ≥50 years of age and have a documented diagnosis of OA in the index knee, based on the American College of Rheumatology (ACR) Criteria for Classification of Idiopathic OA of the knee. Subjects will not be eligible if they have ≥1 pain score reported as 10 on the NRS during the 7 days prior to randomization (Day 1).

For subjects with bilateral knee pain, the more symptomatic knee (i.e., the more painful knee) will be determined by the investigator together with the subject as the index knee during the Screening Visit.

The screening period of the study will include a washout from analgesics and from other drugs taken for pain (i.e nonsteroidal anti-inflammatory drug) that will be followed by a Run-in Period (Day 7 to Day 1) with a total duration of up to 21 days before randomization. Subjects will return to the study site on Day 1 (Baseline), at Weeks 4 (Day 28), 8 (Day 56), 12 (Day 84), 16 (Day 112), 20 (Day 140), 24 (Day 168), and 36 (Day 252) during the double-blind treatment period of 36 weeks to complete the efficacy, safety, and tolerability assessments as applicable. In addition, those approximately 250 subjects who participate in the safety follow up period will return to the site at Week 48 (Day 336). Regular telephone contacts will occur every 2 weeks between scheduled visits during the double-blind treatment and safety follow-up periods to assess the adverse events and to verify treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent for participation in the clinical study.
2. Subject is outpatient of either sex, aged ≥50 years.
3. Subjects with a diagnosis of OA (osteoarthritis) according to the ACR (American College of Rheumatology) criteria.
4. Subject has a radiographic diagnosis (confirmed by a central reader) of knee OA classified Kellgren-Lawrence Grade of 2 or 3 on standing anterior-posterior X-ray of the index knee based on an x ray assessment of both knees available <6 months from Screening or performed during Screening.
5. Subject has a history of knee OA for >6 months (including regular pain and functional impairment) as confirmed by the investigator, based on available written documentation and/or subject reporting.
6. Subject meets the following requirements:

   1. Has a mean score of ≥5 to ≤9 on the 24-hour average daily pain score in the index knee (0-10 Numerical Rating Scale-NRS), where the mean is calculated over all values that are available in the 7 days prior to randomization (Day 1), and it is required that at least 5 pain score values will be available during that period.
   2. Subject has an individual index knee 24-hour average daily pain score ≥1 and ≤9 for all values that are available in the 7 days prior to randomization (Day 1).
7. Subject has rated the pain in the non index knee consistently lower than the pain in the index knee at both the Screening and Baseline Visits in case of bilateral knee OA.
8. Subject, if of childbearing potential, is nonlactating and nonpregnant (has negative serum pregnancy test results at Screening and negative urine pregnancy test result at the start of IP administration prior to dosing).
9. Subject, if female, is either not of childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy, or hysterectomy]) or practicing 1 of the following medically acceptable methods of birth control:

   * Hormonal methods such as oral, implantable, injectable, or transdermal contraceptives for a minimum of 1 full cycle (based on the subject's usual menstrual cycle period) before IP administration.
   * Agrees to abstain from heterosexual intercourse during study participation and to use a highly effective contraceptive (as described above) as backup if they become sexually active during the study. Abstinence is only acceptable if this is the subject's usual lifestyle. Periodic abstinence (calendar, symptothermal, postovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception.
   * Intrauterine device.
   * Double barrier method (condoms, sponge, diaphragm, with spermicidal jellies, or cream).
10. Subject able to understand and follow the study requirements.

Exclusion Criteria:

1. Subject with an allergy or hypersensitivity to the active substance or to any other ingredient of the IP (i.e., chondroitin sulfate tablets or placebo) or has a vegan lifestyle.
2. Subject presenting with lactose intolerance.
3. Subject with ≥1 pain score reported as 10 on the NRS during the 7 days prior to randomization (Day 1).
4. Subject with New York Heart Association Grade III-IV with an ongoing treatment.
5. Subject with severe renal or hepatic impairment (Child-Pugh Stage C) with renal and liver function assessment based on laboratory results.
6. Subject with any other clinically severe or significant uncontrolled concurrent illness.
7. Subject with any other concurrent illness requiring chronic use of analgesics/NSAIDs (nonsteroidal anti-inflammatory drug).
8. Subject has a body mass index ≥40 kg/m2.
9. Subject has predominantly patellofemoral osteoarthritis based on clinical diagnosis and/or x-ray.
10. Subject had surgery of the index knee in the past 6 months (for arthroscopic surgery) or 12 months (for osteotomy or other surgery) or significant injuries in the past 6 months prior to Screening, or has planned knee surgery during the study.
11. Subject with presence of clinical effusion of the knee requiring arthrocentesis or active infection of the index knee.
12. Subject has any important genu varum or valgum >8°(physiological angle including) or any other axial disorder justifying an osteotomy as assessed by central reading.
13. Subject had viscosupplementation, tidal lavage, platelet-rich plasma, or stem cell injection within the last 6 months before Screening.
14. Subject has systemic inflammatory arthropathies (rheumatic disease, inflammatory, infective, or metabolic joint diseases; recurrent clinical chondrocalcinosis; crystal arthropathies; osteo-articular pathologies differing from arthrosis; ochronosis; acromegaly; heritable disorders; or collagen gene mutations), metabolic arthropathies, or Paget's illness.
15. History of acquired or congenital immunodeficiency diseases or positive test results for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus current infection at Screening.
16. Subject has received any of the following:

    * Basic treatment of arthritis with food supplements for joint care (chondroitin sulfate, glucosamine sulfates, diacerein, hyaluronic acid etc.) within the last 3 months.
    * Treatment with oral or parental corticoids during the last month or corticosteroid joint injection within the last 3 months; treatment with inhaled corticosteroids is allowed.
    * Any medication having an influence on pain:

      * NSAIDs (washout period begins ≥5 half-lives of the drug prior to Day 7 and needs to be completed prior to Day 7);
      * Hypnotics, muscle relaxants, anxiolytics, if intake has started <8 days before Screening to be completed prior to Day -7;
      * Use of cannabinoids needs to be stopped ≥2 weeks before the Screening Visit;
      * Acetaminophen or other analgesics (washout period begins ≥5 half-lives of the drug prior to Day 7 and needs to be completed prior to Day -7).
17. Subject has foreseen physiotherapy or alternative medicine (mesotherapy, acupuncture) within the next 12 months (study period).
18. Subject is presenting with clinically relevant psychiatric illness hindering the protocol compliance.
19. Subject is presenting with alcoholism or substance use disorder according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, criteria, or has a positive drug screen result at the Screening or the Baseline Visit. The use of tricyclic antidepressants at low doses for sleep is allowed.
20. Subject has participated in any other clinical study in the month prior to Screening.
21. Subject is noncompliant with eDiary use as determined at the Baseline Visit (i.e., has a compliance <70% throughout the entire Screening Period).

    -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy of once daily treatment-Change in pain (baseline to week-24) in target knee | Week 24
  Change from Baseline to Week 24 in the weekly mean of the average daily pain in the index knee as measured by the numerical rating scale (NRS) (0 10 points where 0 is "no pain" and 10 "the worst pain imaginable")
Safety of the long term treatment-Primary outcome of Safety Follow-up Period from Weeks 36 and 48 with Continued Double-blind Treatment | 48 weeks
  Number of subjects with any AEs, TEAEs, ADRs, and SAEs in Safety Follow-up Period from Weeks 36 and 48 with Continued Double-blind Treatment

SECONDARY OUTCOMES:
Key secondary endpoint of the Double-blind Treatment Period until Week 36. Efficacy of once daily treatment-Change (baseline to week 24) in target knee function | Week 24
  Change from Baseline to Week 24 in Western Ontario and McMaster Universities Arthritis Index (WOMAC) function subscale. WOMAC consists of 24 questions and produces 3 subscale scores for pain (5 questions), stiffness (2 questions), and function (17 questions), and a total score that summarizes overall disability. Only the function subscale will be analyzed for this key secondary endpoint. Each question is scored from 0 to 10 using a standardized 11 point NRS. Each subscale score and the total score will be averaged to provide subscale and total scores between 0 and 10.
Key secondary endpoint of the Double-blind Treatment Period until Week 36. Subject's global evaluation | Week 24
  Subject's global evaluation at Week 24 as measured by Patient Global Impression of Change (PGIC). The PGIC is a self-administered instrument that measures change in subjects' overall improvement with treatment on a scale where 1 = "very much improved" and 7 = "very much worse."
Key secondary endpoint of the Double-blind Treatment Period until Week 36. Durability of the effect (up to week 36) | Week 36
  Durability of effect: change from Baseline to Week 36 in the weekly mean of the average daily pain in the index knee as measured with the Numerical Rating Scale (NRS: 0 10 points where 0 is "no pain" and 10 "the worst pain imaginable")
Safety and tolerability-Double-blind Treatment Period until Week 36. | week 24
  Number of subjects with any AEs, treatment-emergent adverse events (TEAEs), AEs causally related to the investigational product (IP) (adverse drug reactions [ADRs]), and serious adverse events (SAEs)

IPD SHARING:
Plan to Share IPD: No